CLINICAL TRIAL: NCT05929222
Title: An Open-label, Randomized Phase III Trial Comparing Local Radiotherapy Alone or Combined With Obinutuzumab in Early Stage Follicular Lymphoma: the GAZEBO Trial From the Fondazione Italiana Linfomi
Brief Title: Comparison Between Local Radiotherapy Alone or Combined With Obinutuzumab in Early Stage Follicular Lymphoma: the GAZEBO Trial From the Fondazione Italiana Linfomi
Acronym: FIL_GAZEBO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_GAZEBO
Record Dates: First submitted 2023-06-15; First posted 2023-07-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma
Keywords: Lymphoma; Follicular; Immunotherapy; FL; Radiotherapy; Early; Localized; Obinutuzumab; MRD; Minimal residual disease; PET
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma; Neoplasm, Residual | interventions — Radiotherapy; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Active Comparator): Radiotherapy alone
  Interventions: Radiation: Radiotherapy
- Experimental Arm (Experimental): Radiotherapy plus Obinutuzumab
  Interventions: Other: Radiotherapy plus Obinutuzumab

INTERVENTIONS:
Radiation: Radiotherapy — Involved-Site Radiation Therapy 24Gy
  Arms: Standard Arm
Other: Radiotherapy plus Obinutuzumab — Involved-Site Radiation Therapy 24Gy followed by Obinutuzumab 1000mg flat dose 4 doses weekly plus addition 4 doses every 3 weeks
  Arms: Experimental Arm

SUMMARY:
Prospective, multicenter, open label, phase III randomized clinical trial in previously untreated Follicular Lymphoma in early stage. Patients will be randomized to receive Radiotherapy or Radiotherapy plus Obinutuzumab.

DETAILED DESCRIPTION:
Prospective, multicenter, open label, phase III randomized clinical trial in previously untreated Follicular Lymphoma in early stage (I-II non-bulky).

Patients will be randomized to receive:

- Involved-Site Radiation Therapy at standard dose 24Gy - standard arm

OR

- Involved-Site Radiation Therapy at standard dose 24Gy followed by Obinutuzumab 4 infusions weekly + 4 infusions every 3 weeks (8 total doses) - experimental arm

ELIGIBILITY:
Inclusion Criteria:

1. Histological documented diagnosis of Follicular Lymphoma grade I-IIIA as defined in the 2017 edition of World Health Organization (WHO)
2. Ann Arbor Stage IA or IIA (includible in one radiation field), or IE, non-bulky (<7 cm). Stage must be determined by PET/CT scan (Appendix 2)
3. Patients performing PET before surgery can also be enrolled without repeating PET after surgery
4. No previous treatment except for steroid pre-treatment
5. FLIPI < 2, FLIPI2 ≤ 2
6. Age ≥ 18 years
7. Negative bone marrow biopsy
8. Qualitative/quantitative PCR centralized assessment of BCL2/IGH positive cells in peripheral blood (PB), bone marrow (BM).
9. Centralized revision of the lymph node biopsy with FISH for t(14;18)
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
11. At least one site of measurable nodal disease pre-biopsy ≥ 2.0 cm in the longest transverse diameter as determined by CT scan or ultrasonography
12. Adequate renal function defined as follows:

    * Creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)
13. Adequate hepatic function per local laboratory reference range as follows:

    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x UNL
    * Bilirubin ≤1.5 x UNL (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
14. Subject understands and voluntarily signs an informed consent form approved by an Independent National Ethics Committee (NEC), prior to the initiation of any screening or study-specific procedures
15. Subject must be able to adhere to the study visit schedule and other protocol requirements
16. Life expectancy ≥ 3 months
17. Fertility and pregnancy prevention criteria

    * Women must be:

      * postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months)
      * surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
      * completely abstinent (periodic abstinence from intercourse is not permitted) or if sexually active, be practicing a highly effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double barrier method (e.g.: condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization) as local regulations permit, before entry, and must agree to continue to use the same method of contraception throughout the study. They must also be pre-pared to continue birth control measures for at least 18 months after terminating treatment.
    * Women of childbearing potential must have a negative pregnancy test at screening
    * Men with female partners of childbearing potential: men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of study treatment. Men must refrain from donating sperm for the same period
    * Male even if surgically sterilized (i.e., status post vasectomy) must agree to 1 of the following

      * practice effective barrier contraception during the entire study treatment period and through 3 months after the last dose of study drug, or
      * agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner] and withdrawal are not acceptable methods of contraception)

Exclusion Criteria:

1. Histological diagnosis of Follicular lymphoma grade IIIb
2. Staging >II or B symptoms or bulky disease (> 7 cm)
3. Stage II with distant involved sites, not includible in a single radiation field
4. Primary cutaneous follicular lymphoma
5. Known HIV positivity
6. Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RNA on the same sample to confirm the result, if negative, the patient is eligible.
7. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a quantitative HBVDNA test will be performed and if positive the subject will be excluded. Patients with HBcAb positivity and negative HBV DNA should be prophylactically treated with oral Lamivudine (100 mg /day). Note: subjects with serologic evidence of prior vaccination to HBV (i.e., hepatitis B surface (HBs) antigen negative, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
8. Central Nervous System (CNS) involvement with lymphoma
9. Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent
10. Any history of other active malignancies within 3 years prior to study entry, except for adequately treated in situ carcinoma of the cervix uterine, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically resected with curative intent
11. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

    * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
    * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment.
12. If female, the patient is pregnant or breast-feeding
13. Patients participating in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From treatment start up to 33 months (9 months treatment period and 24 months of follow-up)
  Time between the randomization to first documentation of recurrence, progression or death from any cause at 2 years

SECONDARY OUTCOMES:
Complete response rate (CRR) | From therapy start up to end of treatment (9 months)
  Complete response (CR) rate according to the international criteria (Cheson 2014)
Overall response rate (ORR) | From therapy start up to end of treatment (9 months)
  ORR will be defined as the proportion of patients who have a partial or complete response at every treatment phase
Disease Free Survival (DFS) | From post radiotherapy assessment up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Time between the first documentation of Complete Response to any treatment failure, including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of a new treatment without documented progression) or death from any cause
Event Free Survival (EFS) | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Time between the randomization to any treatment failure, including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of a new treatment without documented progression) or death from any cause
Number of patients with Molecular Response at end of treatment | From therapy start up to end of treatment (9 months)
  MRD negativity at end of treatment for positive patients at baseline
Rate of Adverse Events | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Incidence and severity of AEs in both arms according to latest CTCAE criteria
Prognostic and predictive impact of presence/abscence of t(14;18) rearrangement measured by FISH | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Prognostic and predictive impact on PFS in presence or absence of t(14;18) rearrangement measured by FISH
Prognostic role of Minimal Residual Disease by conventional (BCL2/IGH rearrangement by ddPCR) and ctDNA method | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Prognostic role of conventional MRD (BCL2/IGH rearrangement by ddPCR) and of MRD on plasmatic circulating tumour deoxyribonucleic acid (ctDNA) at different time points for PFS and relapse
Prognostic and predictive value of different threshold of metabolic response expressed as SUVmax, MTV and TLG at baseline (PET-0); | At baseline (before therapy start)
  Prognostic and predictive value of different threshold of metabolic response expressed as quantitative PET indexes (QPI) at baseline (PET-0), i.e. SUVmax, MTV and TLG;
Prognostic and predictive role of liquid biopsy by DNA sequencing for lymphoma mutations | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Prognostic and predictive role of liquid biopsy by DNA sequencing for lymphoma mutations at different time points on PFS and relapse
Prognostic and predictive value of radiological markers assessed by Machine Learning tools (pyRadiomics) | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Prognostic and predictive value of radiomic analysis on PFS, assessed on both CT and PET scans by Machine Learning tools (pyRadiomics);
Correlation of MRD results with the radiomics results and clinical outcomes | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Correlation of MRD results with the radiomics results and clinical outcomes
Comparison between genotype at diagnosis and at relapse assessed by RNA sequencing (CIBERSORTx) | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Comparison between genotype at diagnosis and at relapse assessed by RNA sequencing (CIBERSORTx)
Evaluation of liquid biopsy as a tool to identity specific mutations predictive for clonal evolution of lymphoma | From therapy start up to 45 months (9 months treatment phase plus 36 months of follow-up)
  Evaluation of liquid biopsy as a tool to identity specific mutations predictive for clonal evolution of lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pulsoni, MD, Principal Investigator — Ospedale Santa Maria Goretti Latina; Andrea Filippi, MD, Principal Investigator — Università di Pavia-Fondazione IRCCS Policlinico San Matteo
Locations (48):
- Italy (48):
  - Azienda Ospedaliera Nazionale Ss Antonio E Biagio E C Arrigo, SCDU Ematologia, Alessandria
  - AORN San Giuseppe Moscati Avellino, U.O.C. Ematologia e Trapianto Emopoietico, Avellino
  - Centro Di Riferimento Oncologico Di Aviano, S.O.C. Oncologia Medica e dei Tumori Immunocorrelati, Aviano
  - Istituto Tumori Bari Giovanni Paolo II, U.O. di Ematologia e Terapia Cellulare, Bari
  - Ospedale degli Infermi di Biella, SSD Ematologia, Biella
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, U.O. Ematologia, Brescia
  - ARNAS G. Brotzu, SC Ematologia e CTMO, Cagliari
  - Istituto Di Candiolo Fondazione Del Piemonte Per Loncologia IRCCS, Oncologia Medica, Candiolo
  - Istituto Oncologico Veneto, U.O.C. Oncoematologia, Castelfranco Veneto
  - Azienda Ospedaliero Universitaria Policlinico G Rodolico San Marco Di Catania, UOC Ematologia, Catania
  - Azienda Ospedaliera Santa Croce E Carle, S.C. di Ematologia, Cuneo
  - Careggi University Hospital, SOD Ematologia, Florence
  - Ssd Ematologia ASLTO4, S.S.D. Ematologia, Ivrea
  - Ospedale Santa Maria Goretti, SOD Ematologia, Latina
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST S.r.l., Oncoematologia, Meldola
  - Azienda Ospedali Riuniti Papardo-Piemonte, U.O. Ematologia, Messina
  - ASST Grande Ospedale Metropolitano Niguarda, SC Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, S.C. Ematologia e Trapianto Midollo Osseo Allogenico, Milan
  - Ospedale San Raffaele S.r.l., Unitа Linfomi - Dipartimento Oncoematologia, Milan
  - Azienda Ospedaliero Universitaria Di Modena, S.C. Ematologia, Modena
  - Azienda Ospedaliera S Gerardo Di Monza, Ematologia, Monza
  - Azienda Ospedaliera Universitaria Federico II Di Napoli, U.O.C. di Ematologia e Trapianti di Midollo, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore Della Carita, SCDU Ematologia, Novara
  - Istituto Oncologico Veneto, UOC Oncologia 1, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Oncoematologia, Palermo
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, U.O.C. Ematologia, Palermo
  - Fondazione IRCCS Policlinico San Matteo, U.O.C. Ematologia I, Pavia
  - Hospital Santa Maria Della Misericordia, S.C. di Ematologia con TMO, Perugia
  - Azienda Unità Sanitaria Locale Di Piacenza, U.O.Ematologia, Piacenza
  - Azienda Ospedaliero Universitaria Pisana, U.O. Ematologia, Pisa
  - Azienda Unita Sanitaria Locale Della Romagna, U.O.C. Ematologia, Ravenna
  - Azienda USL IRCCS Di Reggio Emilia, S.C. Ematologia, Reggio Emilia
  - Azienda Unita Sanitaria Locale Della Romagna, U.O. di Ematologia, Rimini
  - ASL Roma 1, UOSD Ematologia, Roma
  - Azienda Ospealiero Universitaria Policlinico Umberto I, Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Azienda Ospedaliera S Giovanni Addolorata, UOC Ematologia, Roma
  - Azienda Ospedaliero-Universitaria Sant Andrea, UOC Ematologia, Roma
  - Catholic University Of Sacred Heart, UOC Ematologia e Trapianto di cellule staminali emopoietiche, Roma
  - Fondazione Policlinico Universitario Campus Bio-Medico, UOC di Ematologia e Trapianto di Cellule Staminali, Roma
  - I.F.O. Istituti Fisioterapici Ospitalieri, UOSD Ematologia e Trapianto, Roma
  - Ospedale Di Sassuolo S.p.A., U.O.S.D. di Oncologia, Sassuolo
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Ematologia, Siena
  - Azienda Socio Sanitaria Territoriale Della Valtellina E Dell Alto Lario, Medicina Interna, Sondrio
  - Azienda Ospedaliera S Maria Di Terni, S.C. Oncoematologia, Terni
  - Azienda Unita' Locale Socio Sanitaria N. 2 Marca Trevigiana, S.C di Ematologia, Treviso
  - Azienda Sanitaria Universitaria Friuli Centrale, SOC Clinica Ematologica, Udine
  - Azienda Ospedaliera Ospedale Di Circolo E Fondazione Macchi, U.O.C Ematologia, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona, U.O.C. Ematologia, Verona